CLINICAL TRIAL: NCT00953563
Title: The Mechanism of Action of Unite Biomatrix in Venous Leg Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U0802
Record Dates: First submitted 2009-07-24; First posted 2009-08-06 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Venous Leg Ulcers
Keywords: Venous Leg Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- compression therapy (No Intervention)
- Biologic with compression therapy (Active Comparator)
  Interventions: Device: Unite Biomatrix

INTERVENTIONS:
Device: Unite Biomatrix — collagen based, decellularized equine pericardial dressing for skin surface wounds
  Arms: Biologic with compression therapy

SUMMARY:
The purpose of this study is to assess the mechanism of action of the Unite Biomatrix and compare its performance with the standard of care, compression therapy alone for the treatment of venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* venous ulcer confirmed w/ duplex ultrasound
* ulcer greater than 6 months duration
* post-debridement, the ulcer size must be >5cm2
* at least 18 years old
* ABI is between 0.7 to 1.2 and/or one of the following:

  * TcPO2 > 30mmHg at the ankle
  * Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic)
* able and willing to provide a voluntary written informed consent
* three or fewer ulcers separated by >3.0 cm distance
* able and willing to attend scheduled follow-up visits and study related exams

Exclusion Criteria:

* greater than 20% reduction in wound size during the first 2 weeks of observation with the investigator
* ulcer with exposed bone or tendon
* clinical infection at the studied ulcer site including cellulitis and osteomyelitis
* ulcer of a non-venous insufficiency etiology
* phlebitis or deep leg vein thrombosis in past 30 days
* arterial bypass in previous 30 days
* severe anemia (Hgb<8)
* serum albumin <3.0
* uncompensated congestive heart failure
* renal failure with Creatinine >2.5mg/dl
* rheumatoid arthritis (and other collagen vascular disease), vasculitis, sickle cell disease, HIV
* severe liver disease as defined by treating physician
* uncontrolled diabetes mellitus determined by treating physician
* malignancy at or near the ulcer site
* any condition judged by the PI that would cause the study to be detrimental to the patient
* known allergy to equine derived tissue
* received another investigational device or drug within 30 days of Day 0
* radiation therapy at the wound site
* chemotherapy or immunosuppressive therapy within 30 days of enrollment
* received another allograft, autograft, xenograft within 30 days of the study
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Wound healing pathway markers | baseline, day 0, 3, wk 1, 2

SECONDARY OUTCOMES:
Bacterial Bioburder | baseline, day 0, 3, wk 1, 2

CONTACTS AND LOCATIONS:
Overall Officials: Gerit Mulder, DPM, Principal Investigator — UCSD
Locations (3):
- United States (3):
  - UCSD Medical Center, San Diego, California
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Newbridge Medical Research Corp., Warren General Hosp., Warren, Pennsylvania